CLINICAL TRIAL: NCT01200628
Title: Construction and Validation of a Short Screening Scale for Psychotraumatic Disorders for Inpatients Hospitalized in Surgical Unit Following a Road Traffic Accident
Brief Title: DEPITAC : Short Screening Scale for Psychotraumatic Disorders After Motor Vehicle Accident
Acronym: DEPITAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2006_0632; DGS 2006-0053 (Other: AFSSAPS); PHRC 2006/R1904 (Other: DHOS); 2006-A00180-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2010-03-18; First posted 2010-09-13 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute
Keywords: posttraumatic stress disorder; acute PTSD; PTSD; motor vehicle accident
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Road traffic accident victims: Cohort of patients hospitalized in surgical department after a motor vehicle accident less than 2 weeks
  Interventions: Behavioral: DEPITAC

INTERVENTIONS:
Behavioral: DEPITAC — heteroevaluation scale by a nurse during hospitalization
  Other Names: early screening PTSD scale

SUMMARY:
Posttraumatic stress disorder (PTSD) is a serious and often chronic response to overwhelmingly stressful events as Road Traffic Accident. Moreover PTSD is associated with increased rates of medical morbidity, poor health-related quality of life, and functional impairment. PTSD is prevalent in primary care settings after road traffic accident, where approximately 25% of patients meet diagnostic criteria for the disorder. Despite the development of a number of efficacious behavioral and pharmacological treatments, only a minority of patients with PTSD receive mental health services. PTSD is frequently underrecognized and untreated in Emergency Department and Surgical Unit.

Then, early diagnosis and prevention of PTSD might help to identify patients with PTSD high risk and lead them to benefit of personalized cares. Nevertheless it is not possible (neither useful) to provide psychological cares for each road traffic accident victim.

This is the reason why we think that nurses can help to screen patients who need treatment for PTSD Hypothesis : Recognition of specific clinical or biological signs occurring during road traffic accident victim hospitalization in surgical unit could allow beginning specific treatment using consultation liaison psychiatry.

Early treatment could allow decreasing incidence of psychotraumatic disorders, increasing surgical functional efficacy and improve convalescence programs. The use of a specific questionnaire could help to screen this disorder.

We have created the DEPITAC scale : a short screening questionnaire with 10 items.

This study will be evaluated DEPITAC's 10-item screen for posttraumatic stress disorder (PTSD) for use in surgical or emergency department.

DETAILED DESCRIPTION:
We include 300 road traffic accident victims hospitalized in surgical department (less than 2 weeks). Patients are hospitalized in 5 different hospitals (3 in Lille, 1 in Douai, 1 in Paris). Patients will be evaluated by a short screening questionnaire (DEPITAC's 10 item screen). Patients will be evaluated by phone with a experimented psychologist (Minimal International Neuropsychiatric Interview DSM IV, PTSD Check List symptoms) at 6 weeks, 6 months and 1 year after the accident.

Purposes :

* To evaluate DEPITAC's 10-item screen for posttraumatic stress disorder (PTSD) for use in surgical or emergency department.
* To measure prognosis value of DEPITAC's 10 item screen on acute PTSD (PTSD Check List symptoms (PCLs) 6th week) and late PTSD (PTSD Check List symptoms (PCLs) 6 months and 1 year) or other psychiatric disorder (anxiety, depression or addictive disorder) (Minimal International Neuropsychiatric Interview MINI DSM IV at 6 months and 1 year).
* To compare DEPITAC to Peritraumatic Distress Inventory (PDI) given a the same time.
* To calculate DEPITAC's total score and correlate to the onset of a PTSD at 6 week, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Road traffic accident victims hospitalized in surgical department less than 2 weeks
* Can be called by phone

Exclusion Criteria:

* Patient with a coma for more than 15 minutes
* Patient with a crania traumatism and with loss of consciousness over 15 minutes
* Homeless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include 250 road traffic accident victim hospitalized in surgical department (less than 2 weeks). Patients are hospitalized in 5 different hospitals (3 in Lille, 1 in Douai, 1 in Paris).
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2007-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
DEPITAC's 10 item screen score | six months
  total score of DEPITAC scale

SECONDARY OUTCOMES:
Peritraumatic Distress Inventory (PDI) results | six months / one year
MINI DSM IV results | six months / one year
  Minimal International Neuropsychiatric Interview DSM IV
PTSD Check List symptoms results | six months / one year

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, MD PhD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - University Hospital, Lille, Lille, North
  - General Hospital, Douai, Douai
  - University Hospital, Grenoble, Grenoble
  - Catholic University Hospital of Lille Saint Philibert, Lille
  - Catholic University Hospital of Lille Saint Vincent, Lille
  - Georges Pompidou European Hospital, Paris, Paris

REFERENCES:
- [Derived] Leroy A, Cottencin O, Labreuche J, Mascarel P, De Pourtales MA, Molenda S, Paget V, Lemogne C, Bougerol T, Gregory T, Chantelot C, Demarty AL, Meyer S, Warembourg F, Duhem S, Vaiva G. Four Questions Nurses Can Ask to Predict PTSD 1 Year After a Motor Vehicle Crash. J Trauma Nurs. 2022 Mar-Apr 01;29(2):70-79. doi: 10.1097/JTN.0000000000000638. PMID 35275108